CLINICAL TRIAL: NCT02671487
Title: Mind-Body Skills Groups for Behavioral and Emotional Problems in War-Traumatized Male Adolescents in Gaza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Mind-Body Medicine (Other)
Responsible Party: Principal Investigator, James S. Gordon, M.D., Director, The Center for Mind-Body Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GT-CMBM-002
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Problem Behavior; Aggression; Posttraumatic Stress Disorder
Keywords: Problem Behavior; Aggression; Posttraumatic Stress Disorder; Adolescents
MeSH Terms: conditions — Problem Behavior; Aggression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mind-Body Skills Groups (Experimental): Mind-body skills groups will be administered for 2 hours once a week for 10 weeks and then once a month for 10 months.
  Interventions: Behavioral: Mind-Body Skills Groups
- Wait List Control (No Intervention): No intervention will be administered. Students will have the opportunity to receive the intervention at the end of the study.

INTERVENTIONS:
Behavioral: Mind-Body Skills Groups — Mind-Body Skills groups consist of small groups of about 8-10 participants who learn and practice meditation, guided imagery, breathing techniques, autogenic training, biofeedback, genograms, and self-expression through words, drawings, and movement.
  Arms: Mind-Body Skills Groups

SUMMARY:
The purpose of this study is to determine whether war-traumatize male adolescents with behavioral and emotional problems who participate in mind-body skills groups will have improvement in behavioral and emotional problems, aggression, and posttraumatic stress disorder (PTSD) symptoms, compared to a wait list control group.

DETAILED DESCRIPTION:
Mind-body skills incorporate meditation, guided imagery, breathing techniques, autogenic training, biofeedback, genograms, and self-expression through words, drawings, and movement in a small group setting. These groups have been used in war-traumatize populations in Kosovo, Gaza and the United States. This study will be investigating the effect of the mind-body skills groups on boys with behavioral and emotional problem at a high school in Gaza to determine if there is improvement in behavioral and emotional problems, aggression, and posttraumatic stress disorder. The results will be compared to a control high school with boys who will not be attending mind-body skills groups and who have experienced similar levels of trauma and also have behavioral and emotional problems.

The mind-body skills groups will be held for 2 hours once a week for 10 weeks and then once a month for 10 months. Measures will be taken at baseline, after the 10 week mind-body skills group program and again at 10 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for eligibility for the study will include having a baseline self-reported score of 18 points or higher on the Strengths and Difficulties Questionnaire which indicates high to very high levels of emotional and behavioral problems

Exclusion Criteria:

* None

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire | Change from Baseline to the end of the 10 week program (Post)
  The 25 item Strengths and Difficulties Questionnaire (SDQ) measures behavioral and emotional function. These 25 items are divided into 5 subscales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. The SDQ is scored on a 3 point Likert-type scale with the responses "not true, "somewhat true", and "certainly true". Total SDQ scores include all the subscales except the prosocial scale.
Strengths and Difficulties Questionnaire | Change from the end of the 10 week program (Post) to 10 month-follow up
  The 25 item Strengths and Difficulties Questionnaire (SDQ) measures behavioral and emotional function. These 25 items are divided into 5 subscales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. The SDQ is scored on a 3 point Likert-type scale with the responses "not true, "somewhat true", and "certainly true". Total SDQ scores include all the subscales except the prosocial scale.
Strengths and Difficulties Questionnaire | Change from Baseline to 10 month follow-up after the program ends
  The 25 item Strengths and Difficulties Questionnaire (SDQ) measures behavioral and emotional function. These 25 items are divided into 5 subscales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. The SDQ is scored on a 3 point Likert-type scale with the responses "not true, "somewhat true", and "certainly true". Total SDQ scores include all the subscales except the prosocial scale.

SECONDARY OUTCOMES:
The Aggression Questionnaire | Change from Baseline to the end of the 10 week program (Post)
  Aggression will be measured using the Aggression Questionnaire (AQ) which is a revision of the Buss-Durkee Hostility Inventory that has been widely used to measure aggression. The AQ consists of 34 items scored on a 5 point Likert-type scale with responses ranging from "not at all like me" to "completely like me". The AQ has the following subscales: physical aggression,verbal aggression, anger, hostility, and indirect aggression.
The Aggression Questionnaire | Change from the end of the 10 week program (Post) to 10 month-follow up
  Aggression will be measured using the Aggression Questionnaire (AQ) which is a revision of the Buss-Durkee Hostility Inventory that has been widely used to measure aggression. The AQ consists of 34 items scored on a 5 point Likert-type scale with responses ranging from "not at all like me" to "completely like me". The AQ has the following subscales: physical aggression,verbal aggression, anger, hostility, and indirect aggression.
The Aggression Questionnaire | Change from Baseline to 10 month follow-up after the program ends
  Aggression will be measured using the Aggression Questionnaire (AQ) which is a revision of the Buss-Durkee Hostility Inventory that has been widely used to measure aggression. The AQ consists of 34 items scored on a 5 point Likert-type scale with responses ranging from "not at all like me" to "completely like me". The AQ has the following subscales: physical aggression,verbal aggression, anger, hostility, and indirect aggression.
PTSD Checklist-5 | Change from Baseline to the end of the 10 week program (Post)
  Posttraumatic Stress Disorder (PTSD) Symptoms will be measured using the PTSD Checklist-5 (PCL-5). PCL-5 is a a self-report measure that assesses 20 symptoms of PTSD. The rating scale is 0-4 for each symptom with responses ranging from "Not at all," "A little bit," Moderately," "Quite a bit," to "Extremely."
PTSD Checklist-5 | Change from the end of the 10 week program (Post) to 10 month-follow up
  Posttraumatic Stress Disorder (PTSD) Symptoms will be measured using the PTSD Checklist-5 (PCL-5). PCL-5 is a a self-report measure that assesses 20 symptoms of PTSD. The rating scale is 0-4 for each symptom with responses ranging from "Not at all," "A little bit," Moderately," "Quite a bit," to "Extremely."
PTSD Checklist-5 | Change from Baseline to 10 month follow-up after the program ends
  Posttraumatic Stress Disorder (PTSD) Symptoms will be measured using the PTSD Checklist-5 (PCL-5). PCL-5 is a a self-report measure that assesses 20 symptoms of PTSD. The rating scale is 0-4 for each symptom with responses ranging from "Not at all," "A little bit," Moderately," "Quite a bit," to "Extremely."

CONTACTS AND LOCATIONS:
Overall Officials: Jamil A Atti, MS, Study Director — The Center for Mind-Body Medicine
Locations (1):
- The Center for Mind-Body Medicine, Gaza, Remal Area, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The Center for Mind-Body Medicine Website — http://www.cmbm.org